CLINICAL TRIAL: NCT00906516
Title: A Phase II Protocol for the Use of Neuradiab® Combined With Bevacizumab (Avastin) Therapy in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Neuradiab® Combined With Bevacizumab (Avastin) Therapy in Patients With Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bradmer Pharmaceuticals Inc. (Industry)
Responsible Party: David A. Reardon, MD, The Preston Robert Tisch Brain Tumor Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAD-302
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Brain Tumors
Keywords: Recurrent Glioblastoma multiforme (GBM); Recurrent Brain Tumor; Recurrent Brain Disease; Neuradiab; Avastin; Bevacizumab
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Brain Diseases | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neuradiab in combination with Avastin (Experimental): Patients will be treated following surgical removal of recurrent glioblastoma with a single intracavitary dose of Neuradiab® delivering 44 Gy±10% to the ridge of the surgically created resection cavity followed by therapy with Bevacizumab (Avastin) at a minimum of 30 days after Neuradiab administration.
  Treatment with Bevacizumab will consist of 10mg/kg iv on days 1 and 15 every 28 days. Other chemotherapies (in addition to Avastin) will be permitted based on most current clinical practice and clinical evaluation of the patient.
  Interventions: Drug: Neuradiab in combination with Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Neuradiab in combination with Bevacizumab (Avastin) — Patients will be treated following surgical removal of recurrent glioblastoma with a single intracavitary dose of Neuradiab® delivering 44 Gy±10% to the ridge of the surgically created resection cavity followed by therapy with Bevacizumab (Avastin) at a minimum of 30 days after Neuradiab administration.
  Treatment with Bevacizumab will consist of 10mg/kg iv on days 1 and 15 every 28 days. Other chemotherapies (in addition to Avastin) will be permitted based on most current clinical practice and clinical evaluation of the patient.
  Other Names: 131I-labeled anti-tenascin murine monoclonal antibody;; Bevacizumab

SUMMARY:
Bradmer Pharmaceuticals, Inc. (Bradmer) is requesting approval to study the safety of Neuradiab® when combined with Bevacizumab (Avastin) therapy given at a minimum of 30 days after Neuradiab administration in patients with a first or second recurrence of glioblastoma multiforme (GBM), in an attempt to manage life threatening recurrence of Grade IV malignant glioma.

DETAILED DESCRIPTION:
At present there are no satisfactory therapies for these patients with recurrent GBM and the practitioner is left with best effort combination therapy for this disease. At present a number of chemotherapeutic agents, including nitrosoureas, carboplatin, bevacizumab, etoposide, irinotecan, and imatinib, have been used as salvage therapy either alone or in combination. Additional trials with a variety of agents are underway, but preliminary results from single-agent studies have been disappointing. Currently, only nitrosoureas (lomustine and carmustine), including Gliadel® Wafer (carmustine) as adjunct to surgery, are approved for use in previously treated GBM. At present the treatment of recurrent disease with any available agent results in median survival in the ranges of 22-44 weeks. The historical data from previous human exposure with Neuradiab is highly suggestive of a benefit to patient survival.

Since Neuradiab® has shown promising efficacy in patients with recurrent disease with acceptable risk-benefit ratio, and since there is no substantial survival benefit from currently available agents used to treat this patient population, Neuradiab® is being proposed as an experimental alternative to recurrent GBM patients under a Single-Center Phase II Trial. Recurrent GBM is a serious and immediately life-threatening disease, for which there is no comparable or satisfactory alternative drug or other therapy available to treat that stage of the disease. Overall, survival data indicate a need for more effective treatments for recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

* Previous histopathology confirmed diagnosis of (World Health Organization [WHO] grade IV astrocytoma; (http://rad.usuhs.mil/rad/who/who2b.html)
* Patients with recurrent disease presenting as a supratentorial unifocal lesion seen on magnetic resonance imaging (MRI) suspicious for glioblastoma multiforme will be considered as long as:

  1. Patient is eligible for or has undergone a gross total surgical resection of the tumor mass with a residual ridge ≤ 1cm
  2. A post-operative MRI will be obtained within 72 hours of resection and must show an adequate resection defined by ≤ 1 cm enhancement.
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are postoperative grade 1.
* Age ≥ 18 years of age at the time of study entry.
* Karnofsky Performance Status ≥ 70%.
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Patient must be HAMA negative prior to study entry
* Able to tolerate standard post operative management for GBM debulking including corticosteroid therapy
* An interval of at least 30 days from prior chemotherapy (6 weeks for nitrosoureas) or investigational agent unless the patient has recovered from all anticipated toxicities associated with that therapy
* Women of childbearing potential must have a negative pregnancy test (serum or urine).
* The patient must agree to use an effective contraceptive method
* Patient must give written informed consent prior to any study-specific procedures being implemented

Exclusion Criteria:

* Infratentorial tumor, tumor with subependymal spread, multifocal tumor, tumor with ventricular communication, intraventricular tumor or tumor which is within one gyrus (approximately 1cm) of the motor/sensory strip, either of the speech centers, or exceeds beyond the cranial vault.
* Severe, active comorbidity, including any of the following:

  1. Unstable angina and/or congestive heart failure requiring hospitalization
  2. Transmural myocardial infarction within the last 6 months
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study entry
  4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study entry
  5. Known hepatic insufficiency resulting in clinical jaundice (excluding Gilbert's syndrome) and/or coagulation defects
  6. Known AIDS based upon current CDC definition
  7. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
  8. Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
* History of severe allergic reaction to contrast media.
* Any serious medical condition or psychiatric illness unresponsive to medical intervention.
* Prior malignancy if active treatment was required during the previous 3 years (except for adequately treated basal cell or squamous cell skin cancer and prior GBM)
* Known hypersensitivity to murine proteins.
* Inability to undergo an MRI.
* Patient has been treated with any anti-angiogenic therapy within 30 days prior to study entry
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The safety of Neuradiab® when followed by Avastin therapy will be assessed based on Investigator reported symptomatic toxicity findings on physical exam, and Adverse Events. | One year

SECONDARY OUTCOMES:
Overall survival (OS). Data will be reported based on a dataset of 60 patients. | One year
Time to progression (TTP). Data will be reported based on a dataset of 60 patients. | One year

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — The Preston Robert Tisch Brain Tumor Center
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

REFERENCES:
- See also: Sponsor Web Site — http://www.bradmerpharma.com